CLINICAL TRIAL: NCT07101263
Title: Hydrolyzed Whey for Blood Lipid Control
Brief Title: Whey Protein Comparisons for Blood Lipid Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medinutra LLC (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Robert DiSilvestro, President, Medinutra LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Medinutra002
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cholesterol
Keywords: Cholesterol; Whey; inflammation; Moderately elevated cholesterol; High end normal cholesterol
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard whey (Placebo Comparator): A standard whey protein is consumed daily for 6 weeks
  Interventions: Dietary Supplement: Standard whey
- Hydrolyzed whey (Experimental): A hydrolyzed whey protein is consumed daily for 6 weeks
  Interventions: Dietary Supplement: Hydrolyzed whey

INTERVENTIONS:
Dietary Supplement: Standard whey — A typical whey protein is given that differs in chemical structure from the atypical whey protein used in the experimental group
  Arms: Standard whey
Dietary Supplement: Hydrolyzed whey — This type of whey has different chemical structure from typical wheys such as that used in this nstudy's control group
  Arms: Hydrolyzed whey

SUMMARY:
The goal of this clinical trial is to learn if hydrolyzed whey protein can help serum cholesterol stay in normal range in adults. As a side inquiry, a few blood measures will be taken that are relevant to low level inflammation. The main questions the study aims to answer are:

* Will hydrolyzed whey lower serum cholesterol readings in adults with starting values in the upper end of normal to the lower end of elevated?
* Will the hydrolyzed whey affect a general measure of inflammation and two measures of indirect relevance to inflammation?

Researchers will compare hydrolyzed whey to a conventional whey (a control protein not expected to affect serum cholesterol readings) to see if the hydrolyzed whey lowers serum cholesterol.

Participants will:

* Drink one protein beverage every day for 6 weeks;
* Go to a LabCorp facility for a blood draw before and after the 6 weeks.

DETAILED DESCRIPTION:
Background. According to the American Medical Association and the Centers for Disease Control, nearly 94 million adults over the age of 20 have what could be considered borderline high cholesterol. Most of these people don't take drugs to lower cholesterol. Therefore, this group of people represent a target for other approaches to lowering cholesterol readings. This group can include people in the high end of acceptable range since they can run the risk of getting into borderline high readings. A nutritional product could be part of a plan to keep cholesterol readings in the normal range.

Whey protein could comprise such a product. This protein gets used in many protein powders, ready-to-drink beverages and bars. However, whey does not have a simple and consistent record for lowering cholesterol readings. Even with the studies giving positive results, only indirect effects may occur. This can happen by whey replacing fat and high glycemic index carbohydrate foods, or by impacting satiety.

In contrast, this project tests the proposition that certain versions of hydrolyzed whey can directly exert a modest but useful action on cholesterol readings. The applicant has found this in a small unpublished study in older exercisers. In addition, a retracted study has shown that in people with pre-hypertension or moderate hypertension, hydrolyzed whey can reduce total and LDL cholesterol readings. A decrease of 29 mg/dL for total cholesterol despite only moderately high starting cholesterol values).

Although this data is useful, it is based only an unpublished study and a retracted paper. Also, the two populations studied were somewhat narrow. Thus, a new study is now going to be done in a fairly broad population. Positive results in this and possible subsequent research could be applied to products quickly since no drug claim is needed. The Dietary Supplement and Education Act (DSHEA) allows for structure function claims of helping maintain blood lipids in the normal range.

As a side note, hydrolyzed whey protein could also reduce low level general inflammation. This process, which falls below what's seen with inflammatory diseases or injury, can raise the risk for many long term health problems. Drugs are not generally employed to minimize this type of inflammation. So, as with moderately high TG readings, relatively safe and inexpensive non-drug alternatives can be sought (including nutritional supplements).

Methods. Subjects will be adult males and females aged 21-59 that lack unstable health problems that can affect cholesterol or systemic inflammation readings. Subjects in this project will have starting total cholesterol reading of 190-225 mg/dL. Initially, this eligibility will be based on eligibility questionnaire. However, if the initial blood draw finds cholesterol readings outside the range, subjects will be excluded and replaced. Other discontinuations will be for a subject's decision or a change in health or medication disclosed by the subject to Medinutra. For these discontinuations, subjects will not be replaced (see next section).

For 6 weeks, subjects will take one of the following orally as one serving/day (up to16 people/group):

Hydrolyzed whey (Hilmar) 25g protein/day Whey protein isolate (Hilmar) 25g protein/day

Blood will be drawn and analyzed at a LabCorp facility. The blood draw site will vary according to the location where each subject lives. Neither Labcorp nor the study subjects will not know the assigned protein identity. Thus, this will be double blinded and randomized in terms of the participants and analyzers

Measures will consist of blood lipids and three measures directly or indirectly related to low level inflammation. For each measure, for each of the 2 treatment groups, pre- and post-treatment values will be compared by paired t-test. In addition, the changes in values for each group will be compared to each group by unpaired t-test. For non-normal distribution, nonparametric tests can be used. Significance for all analysis is set at p < 0.05.

Subject numbers and power calculation. Subject number will be 36/group. For a power calculation, for hydrolyzed whey alone, the 7% change in total cholesterol from the applicant pilot study is used as the minimal desired change. The comparison protein is assumed to have about a 0% change. The variation is set at 4.8%. This produces a power value of 0.95 with a two way p value of 0.01 for 34 subjects per group. An extra 2 subjects per group will be added in case of dropouts. Dropouts are not expected to happen at a high rate since only two trips are required to a site, drinking a protein beverage is not overly hard, and subjects will not be able to tell if an effect is occurring during the study. In the last regard, this study does not resemble something like osteoarthritis research where non-improving pain can make a person drop out.

Safety considerations. Ingestion of any type of beverage as well as having blood draws have some risks, but major risks are not common. The main concern of this study is allergies to whey protein. If someone has allergies to whey, then allergies to milk proteins would also be expected. Therefore, if someone has had milk allergies, then they should not participate in the study. Some people have claimed that allergies to whey can show up even if milk protein allergies exist, but this contention lacks confirmation. However, if a person has ever had any discomfort after consuming whey, then they should not participate.

ELIGIBILITY:
Inclusion Criteria:

* Cholesterol reading of 190 to 225 mg/dL
* Age 21-59 years old

Exclusion Criteria:

* Uncontrolled diabetes
* Hypothyroidism or other hormonal problems that have not stabilized
* Any liver diseases being actively treated
* Cancer
* Renal dialysis use
* Rheumatoid arthritis and related issues like lupus
* Inflammatory bowel disease
* Smoking
* Following a very restrictive diet
* Low blood pressure
* Statin drug use
* Having more than 5 alcoholic drinks per week
* Extreme obesity (BMI over 37)
* Pregnancy or lactation
* Allergies to milk protein
* History of discomfort after consuming whey protein

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Serum cholesterol | 6 weeks
  Serum total and LDL cholesterol (mg/dL) will be assessed

SECONDARY OUTCOMES:
Other Blood Lipids | 6 weeks
  Serum HDL cholesterol and triglycerides (mg/dL) will be assessed, but mean values are not expected to change in either group
Inflammation markers | 6 weeks
  As a secondary consideration, this study will assess 3 blood measures relevant to low level inflammation: serum c reactive protein (mg/dL), serum alanine aminotransferase (ALT-Units/L), and whole blood glutathione (mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Medinutra LLC, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pins JJ, Keenan JM. Effects of whey peptides on cardiovascular disease risk factors. J Clin Hypertens (Greenwich). 2006 Nov;8(11):775-82. PMID 17086017
- See also: The American Medical Association and the Centers for Disease Control reported that nearly 94 million adults over the age of 20 have what could be considered borderline high cholesterol — https://www.ama-assn.org/delivering-care/hypertension/what-doctors-wish-patients-knew-about-high-cholesterol